CLINICAL TRIAL: NCT04939233
Title: Robotic Hand Orthosis Providing Grasp Assistance for Patients With Brachial Plexus Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 19-330; 1R21HD095027-01A1 (NIH)
Record Dates: First submitted 2021-05-28; First posted 2021-06-25 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Brachial Plexus Injury

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Exoskeleton Glove (Experimental): Perform a feasibility trial of the robotic orthosis device by providing it to a small cohort of adult patients suffering from paralysis due to a brachial plexus injury.
  Interventions: Device: Exoskeleton glove

INTERVENTIONS:
Device: Exoskeleton glove — A robotic hand orthosis (exoskeleton glove) will have been developed that is able to naturalistically bend the finger joints of the individuals based on intuitive voice commands

SUMMARY:
The proposed research, the development of an innovative robotic hand orthosis with intelligent grasping control, is relevant to public health as it will restore a large measure of functionality to the paralyzed hand of a person who has suffered a brachial plexus injury. The proposed orthosis will utilize novel technology that will result in a device that is compact, portable, dexterous, and intuitively controllable while overcoming the disadvantages of previously developed orthoses that rendered them difficult to use. The restoration of functionality to ones hands will significantly improve their quality of life as well as their ability to again participate in the workforce and complete dexterous activities in their daily lives.

DETAILED DESCRIPTION:
The overall objective of this research is to design, fabricate, integrate, and test a lightweight and portable robotic hand orthosis intended to restore hand functionality through fully controllable individual finger actuation. This objective is based on the hypothesis that use of such a robotic hand orthosis will result in significant improvement of hand ability for adults with brachial plexus injury, as evaluated through the Southampton Hand Assessment Procedure (SHAP).

To achieve this, several novel design aspects are incorporated. The use of miniature linear actuators and lightweight materials allows for the motors and sensors to all mount atop the dorsum of the hand, and eliminate the need for bulky external actuation units. In addition, the actuators have inbuilt force sensing capabilities to provide feedback on the force being applied to each individual finger, even before contact is made with a grasped object. Furthermore, wrist flexion/extension is powered, resulting in a more realistic grasping paradigm than is commonly found in robotic orthoses. Moreover, an intuitive control system will be designed in order to fully capitalize on the controllability of each finger, allowing for varied grasp geometries and motions.

A summary of the specific aims of this study are:

Design and prototype the robotic hand orthosis with the goal of creating a uniquely dexterous, lightweight and portable device. In addition, the control methodologies required to exploit the full capabilities of the orthosis will be designed. This will result in the development of an experimental research platform to determine the viability of the design and hypothesis.

Perform a feasibility trial of the robotic orthosis device by providing it to a small cohort of adult patients suffering from paralysis due to a brachial plexus injury. The patients will be assessed via the SHAP, and their respective scores both with and without the orthosis will be evaluated to determine their level of improvement in dexterity and function.

ELIGIBILITY:
Inclusion Criteria:

* Brachial plexus injury to the right upper extremity
* 18 - 69 y/o with pan plexus injuries
* Lower root injuries (C7, C8, T1)

Exclusion Criteria:

* No significant hand/wrist contractures or associated deformities which would affect participation
* No open wounds in affected hand or wrist
* Able to provide consent for treatment and follow general directions
* Only right-hand involved individuals will be considered, as the orthosis prototypes will be designed for right hand use only at this stage of the research

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cesar J Bravo, MD, Principal Investigator — Carilion Clinic Ortho Surgeon
Locations (1):
- Carilion Clinic Institute for Orthopaedics and Neurosciences, Roanoke, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exoskeleton Glove
Started | 3 (Four clinical trials involving three participants)
Completed | 3 (Four clinical trials involving three participants)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Exoskeleton Glove
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (0.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Successful Grasp Trials Per Participant Using Robotic Hand Orthosis
Description: Southampton Hand Assessment Procedure (SHAP) Construct Measured: Functional hand performance based on prehensile and Activities of Daily Living (ADL) tasks.
  Structure: 6 Abstract Object Tasks (grip patterns). The five most used grasp types in ADLs were selected for the experiments, which include cylinder grasp, sphere grasp, tip grasp, tripod grasp, and lateral grasp. We selected ten objects that belong to different grasp types for the experiments. Each object was grasped for five times by each participant.
  Scoring: Successful vs unsuccessful grasps with 10 different objects Interpretation: Successful grasps with 10 different objects
Time Frame: The total expected time for the study is about 2 hours.
Measure: Mean (Full Range); unit: Number of successful grabs of an object
Arm/Group | Exoskeleton Glove
Number analyzed (Participants) | 3
Number of successful grabs of an object | 13.2 [0 to 15]

ADVERSE EVENTS:
Time Frame: 1 day
Description: The only potential risk is slight discomfort while wearing the device. The device itself will be designed such that it cannot violate normal human ranges of motion in the hand and is free of potential pinch points. Furthermore, the devices motion can be immediately stopped if necessary.
Arm/Group | Exoskeleton Glove
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT04939233/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT04939233/ICF_001.pdf